CLINICAL TRIAL: NCT06144957
Title: SLC13A5 Deficiency: A Prospective Natural History Study - United States Only
Brief Title: SLC13A5 Deficiency Natural History Study - United States Only
Status: Enrolling by invitation | Type: Observational
Sponsor: TESS Research Foundation (Other)
Collaborators: Stanford University (Other); Brown University (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SLC13A5USNHS
Record Dates: First submitted 2022-01-07; First posted 2023-11-22 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-11

CONDITIONS: Citrate Transporter Deficiency; Epilepsy; Rare Diseases; Movement Disorders; Genetic Disorder; SLC13A5 Deficiency; EIEE25; Kohlschutter-Tonz Syndrome (Non-ROGDI); Citrate Transporter Disorder; DEE25
Keywords: Epilepsy; Rare Disease; Movement Disorders; Genetic Disorder; Citrate Transporter Disorder; SLC13A5 Deficiency; EIEE25; Neonatal seizures; autosomal recessive; DEE25
MeSH Terms: conditions — Epilepsy; Rare Diseases; Movement Disorders; Genetic Diseases, Inborn; Kohlschutter Tonz syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Urine of the Patients and/or their parents will be collected for lab analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
SLC13A5 deficiency (Citrate Transporter Disorder, EIEE 25) is a rare genetic disorder with neurodevelopmental delays and seizure onset in the first few days of life. This natural history study is designed to address the lack of understanding of disease progression. Additionally it will identify clinical and biomarker endpoints for use in future clinical trials.

DETAILED DESCRIPTION:
This is a longitudinal observational study of the natural history of SLC13A5 deficiency for up to 2 years. This study does not involve any therapeutic intervention. The study includes in-person clinical assessments and laboratory analyses including standardized clinical evaluations, neurocognitive and quality of life scales, video movement rating scale, laboratory measurements of blood and urine, EEG capturing wake and sleep, EKG. Additionally, remote assessments in 1st year (every 3 months) and 2nd year (every 4 months) of enrollment will be made and caregiver will be asked to keep a seizure diary for the duration of the study. Personnel having expertise to comprehensively evaluate biological pathways that are perturbed by SLC13A5 deficiency will analyze the collected data. Improved understanding of disease pathogenesis will guide therapeutics and reveal clinical and biomarker endpoints for use in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Parent(s)/legal representative and/or patient must be willing and able to give informed consent/assent for participation in the study.
2. Males and females of any age are eligible for this study
3. Suspected or confirmed diagnosis of SLC135 deficiency with genetic variants in both SLC13A5 alleles and consistent clinical characteristics. Variants of uncertain significance in one or both alleles are acceptable if deemed good candidates by participant's primary geneticist or neurologist and study personnel.
4. Participant and caregiver must be willing to provide clinical data, participate in standardized assessments, and provide biological samples.
5. Willingness to travel to one of the three sites annually is favored, but not required.

Exclusion Criteria:

1. The presence of a second, confirmed disorder, genetic or otherwise, affecting neurodevelopment or with other overlapping symptoms of SLC13A5 deficiency.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of children, adolescents, and adults with suspected or confirmed diagnosis of SLC13A5 Deficiency and consistent clinical characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Detailed phenotyping of the clinical course of SLC13A5 deficiency over time: general evaluations | Up to 24 months
  Conducted in patients with SLC13A5 deficiency: general appearance, HEENT, neck, chest and lungs, cardiovascular, abdomen, genitourinary, rectal, musculoskeletal, lymph nodes, extremities/skin, mental status (alertness, interaction, language (EXP) (REC)), emotional affect (calm, smiling, laughing, anxious, frowning, crying, irritable, screaming).
  As much information as available will also be collected from existing medical records including clinical evaluations, imaging studies and neuropsychological and motor function evaluations.
Detailed phenotyping of the clinical course of SLC13A5 deficiency over time: vitals and biometrics evaluations | Up to 24 months
  Conducted in patients with SLC13A5 deficiency: height (cm), weight (kg), blood pressure (systolic and diastolic), temperature (c), heart rate (beats/minute), respiratory rate (breaths/minute), and head circumference (cm).
  As much information as available will also be collected from existing medical records including clinical evaluations, imaging studies and neuropsychological and motor function evaluations.
Detailed phenotyping of the clinical course of SLC13A5 deficiency over time: neurologic evaluation | Up to 24 months
  Conducted in patients with SLC13A5 deficiency: motor, motor stability, muscle bulk, paresis, sensation, reflexes, coordination, gait, and autonomic.
  As much information as available will also be collected from existing medical records including clinical evaluations, imaging studies and neuropsychological and motor function evaluations.
Detailed phenotyping of the clinical course of SLC13A5 deficiency over time: dental evaluations | Up to 24 months
  Conducted in patients with SLC13A5 deficiency: baseline pain assessment from a scale of 0-10 (0 being no pain and 10 being highest pain), temperature pain assessment for cold from a scale of 0-10 (0 being no pain and 10 being highest pain), temperate pain assessment for hot from a scale of 0-10 (0 being no pain and 10 being highest pain), toothpaste use (type and frequency), and Fluoride treatments.
  As much information as available will also be collected from existing medical records including clinical evaluations, imaging studies and neuropsychological and motor function evaluations.
Detailed phenotyping of the clinical course of SLC13A5 deficiency over time: clinical and research laboratory studies | Up to 24 months
  Conducted in patients with SLC13A5 deficiency:
  Clinical: ammonia, amylase, CKMB, GGT, lactate, lipase, PT/PTT, vitamin d 25-oh, CBC with differential, comprehensive MET panel, lipid panel with calculated LDL, and urine studies (calcium/creatinine ratio, spot ph, spot citrate concentration, citrate/creatinine ratio).
  Research: Citrate and metabolomics.
  As much information as available will also be collected from existing medical records including clinical evaluations, imaging studies and neuropsychological and motor function evaluations.
Detailed phenotyping of the clinical course of SLC13A5 deficiency over time: electroencephalogram (EEG) | Up to 24 months
  Conducted in patients with SLC13A5 deficiency: looking at the duration of EEG, if they are captured awake or asleep, and if it is abnormal.
  As much information as available will also be collected from existing medical records including clinical evaluations, imaging studies and neuropsychological and motor function evaluations.
Detailed phenotyping of the clinical course of SLC13A5 deficiency over time: scoring of movement disorder and SLC13A5 deficiency symptom scales | Up to 24 months
  Conducted in patients with SLC13A5 deficiency: using scale titled "Movement Exam for SLC13A5 Natural History Study". Assessing typical gait, standing in natural position, sitting on chair, head control, attempt to vocalize, speech quality, speech content, ability to grab items, and ability to draw. Symptom scales consist of chorea, dystonia, ataxia, myoclonus, tremor, hypokinetic-rigid syndrome, and tic.
  As much information as available will also be collected from existing medical records including clinical evaluations, imaging studies and neuropsychological and motor function evaluations.
Neurodevelopmental profile of SLC13A5 deficiency as measured using Mullen Scales of Early Learning | Up to 24 months
  Consists of a gross-motor scale and four cognitive scales: visual reception, fine motor, receptive language, and expressive language. T-Scores (mean of 50 and a standard deviation of 10) are given for individual scales, and an optional Early Learning Composite standard score (mean of 100 and a standard deviation of 15) serves as an overall estimate of cognitive functioning. This is based on child's age and there are no higher or lower scores that indicate a better or worse outcome.
  Developmental assessment at baseline and longitudinally, if age and ability-appropriate.
Neurodevelopmental profile of SLC13A5 deficiency as measured using the Peabody Developmental Motor Scales-2 | Up to 24 months
  Six subtests that measure motor ability in children: reflexes, stationary, locomotion, object manipulation, grasping, and visual motor integration. The Peabody has quotients that measure a child's motor ability: gross motor quotient, fine motor quotient, total motor quotient. This is based on child's age and there are no higher or lower scores that indicate a better or worse outcome.
  Developmental assessment at baseline and longitudinally, if age and ability-appropriate.
Neurodevelopmental profile of SLC13A5 deficiency as measured using the Vineland-III Adaptive Behavior Scale | Up to 24 months
  Vineland is a semi-structured interview that assesses adaptive behavior in several domains, summarized by the Adaptive Behavior Composite (ABC) standard score. ABC standard scores may range from 20 to 160, with a population mean of 100 and a standard deviation of 15. There are no higher or lower scores that indicate a better or worse outcome.
  Developmental assessment at baseline and longitudinally, if age and ability-appropriate. Additionally, Vineland-III Adaptive Behavior Scale questionnaire will be included in the remote assessment interview.
Seizure burden and semiology as measured using the Seizure Global Impression of Change | Up to 24 months
  Assessing the status of the patient's overall condition using a scale ranging from very much improved, much improved, slightly improved, no change, slightly worse, much worse, very much worse. Assessing the average number of participants' seizures on a scale of decreased, stayed the same, increased. Assessing the average duration of the participants' seizures on a scale of decreased, stayed the same, increased.
  Caregiver will be asked to maintain a seizure diary throughout the study and seizure burden will be assessed at in-person and remote assessments.

SECONDARY OUTCOMES:
Participant quality of life as measured through the Pediatric Quality of Life Inventory (PedsQL) Family Impact | Up to 24 months
  The PedsQL Family Impact Module measures parent self-reported physical, emotional, social, and cognitive functioning, communication, and worry. The Module also measures parent-reported family daily activities and family relationships.
  Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher scores indicate better functioning (less negative impact). Scale Scores are computed as the sum of the items divided by the number of items answered (this accounts for missing data).
  Quality of life will be evaluated at baseline and longitudinally.
Participant quality of life as measured through the Pediatric Quality of Life Inventory (PedsQL) Caregiver Epilepsy Module | Up to 24 months
  The PedsQL Epilepsy Module is a 29-item measure with five scales: Impact, Cognitive, Sleep, Executive Function, and Mood/Behavior.
  Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher scores indicate better functioning (less negative impact). Scale Scores are computed as the sum of the items divided by the number of items answered (this accounts for missing data).
  Quality of life will be evaluated at baseline and longitudinally.
Participant sleep disturbances as measured through the Sleep Disturbances Scale for Children (SDSC) | Up to 24 months
  Consisting of 26 Likert-type items, the SDSC was designed both to evaluate specific sleep disorders in children, and to provide an overall measure of sleep disturbance suitable for use in clinical screening and research.
  Higher scores indicate more acute sleep disturbances. To obtain results, scores are tallied for each of the six sleep-disorder categories, and an overall score is calculated.
  The sleep disturbances will be evaluated at baseline and longitudinally.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda E Porter, MD, PhD, Principal Investigator — Stanford University; Kimberly Goodspeed, MD, PhD, Principal Investigator — University of Texas Southwestern Dallas; Judy Liu, MD, PhD, Principal Investigator — Brown University
Locations (3):
- United States (3):
  - Lucille Packard Children's Hospital, Stanford University, Palo Alto, California
  - Brown University, Providence, Rhode Island
  - University of Texas Southwestern Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The study data will be retained in the study-specific REDCap data base housed at redcap.stanford.edu. Researchers and clinicians with academic interest in SLC13A5 deficiency may be provided access to data obtained through this study. Any data shared outside of Stanford University will be done so in a coded fashion with no protected health information included and with the execution of all applicable agreements or ongoing collaborations as approved.

REFERENCES:
- [Background] Thevenon J, Milh M, Feillet F, St-Onge J, Duffourd Y, Juge C, Roubertie A, Heron D, Mignot C, Raffo E, Isidor B, Wahlen S, Sanlaville D, Villeneuve N, Darmency-Stamboul V, Toutain A, Lefebvre M, Chouchane M, Huet F, Lafon A, de Saint Martin A, Lesca G, El Chehadeh S, Thauvin-Robinet C, Masurel-Paulet A, Odent S, Villard L, Philippe C, Faivre L, Riviere JB. Mutations in SLC13A5 cause autosomal-recessive epileptic encephalopathy with seizure onset in the first days of life. Am J Hum Genet. 2014 Jul 3;95(1):113-20. doi: 10.1016/j.ajhg.2014.06.006. PMID 24995870
- [Background] Hardies K, de Kovel CG, Weckhuysen S, Asselbergh B, Geuens T, Deconinck T, Azmi A, May P, Brilstra E, Becker F, Barisic N, Craiu D, Braun KP, Lal D, Thiele H, Schubert J, Weber Y, van 't Slot R, Nurnberg P, Balling R, Timmerman V, Lerche H, Maudsley S, Helbig I, Suls A, Koeleman BP, De Jonghe P; autosomal recessive working group of the EuroEPINOMICS RES Consortium. Recessive mutations in SLC13A5 result in a loss of citrate transport and cause neonatal epilepsy, developmental delay and teeth hypoplasia. Brain. 2015 Nov;138(Pt 11):3238-50. doi: 10.1093/brain/awv263. Epub 2015 Sep 17. PMID 26384929
- [Background] Klotz J, Porter BE, Colas C, Schlessinger A, Pajor AM. Mutations in the Na(+)/citrate cotransporter NaCT (SLC13A5) in pediatric patients with epilepsy and developmental delay. Mol Med. 2016 May 26;22:310-21. doi: 10.2119/molmed.2016.00077. PMID 27261973
- [Background] Selch S, Chafai A, Sticht H, Birkenfeld AL, Fromm MF, Konig J. Analysis of naturally occurring mutations in the human uptake transporter NaCT important for bone and brain development and energy metabolism. Sci Rep. 2018 Jul 27;8(1):11330. doi: 10.1038/s41598-018-29547-8. PMID 30054523
- [Background] Bainbridge MN, Cooney E, Miller M, Kennedy AD, Wulff JE, Donti T, Jhangiani SN, Gibbs RA, Elsea SH, Porter BE, Graham BH. Analyses of SLC13A5-epilepsy patients reveal perturbations of TCA cycle. Mol Genet Metab. 2017 Aug;121(4):314-319. doi: 10.1016/j.ymgme.2017.06.009. Epub 2017 Jun 24. PMID 28673551
- [Background] Weeke LC, Brilstra E, Braun KP, Zonneveld-Huijssoon E, Salomons GS, Koeleman BP, van Gassen KL, van Straaten HL, Craiu D, de Vries LS. Punctate white matter lesions in full-term infants with neonatal seizures associated with SLC13A5 mutations. Eur J Paediatr Neurol. 2017 Mar;21(2):396-403. doi: 10.1016/j.ejpn.2016.11.002. Epub 2016 Nov 19. PMID 27913086
- [Background] Irizarry AR, Yan G, Zeng Q, Lucchesi J, Hamang MJ, Ma YL, Rong JX. Defective enamel and bone development in sodium-dependent citrate transporter (NaCT) Slc13a5 deficient mice. PLoS One. 2017 Apr 13;12(4):e0175465. doi: 10.1371/journal.pone.0175465. eCollection 2017. PMID 28406943
- [Background] Schossig A, Bloch-Zupan A, Lussi A, Wolf NI, Raskin S, Cohen M, Giuliano F, Jurgens J, Krabichler B, Koolen DA, de Macena Sobreira NL, Maurer E, Muller-Bolla M, Penzien J, Zschocke J, Kapferer-Seebacher I. SLC13A5 is the second gene associated with Kohlschutter-Tonz syndrome. J Med Genet. 2017 Jan;54(1):54-62. doi: 10.1136/jmedgenet-2016-103988. Epub 2016 Sep 6. PMID 27600704